CLINICAL TRIAL: NCT06758674
Title: The Effect of the Training Program Given to Bedridden Patients At Home to Prevent Pressure Ulcer Development on Pressure Ulcer Formation
Brief Title: The Effect of an Training Program for the Prevention of Pressure Ulcers in Bedridden Patients At Home
Acronym: no acronym
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ozcan, Nurse, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IKCU-SBF-AO-01; 2024-TYL-SABE-0027 (Other Grant/Funding Number: Izmir Katip Celebi University Scientific Research (Master Thesis) Project)
Record Dates: First submitted 2024-12-27; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Pressure Ulcer Prevention
Keywords: pressure ulcer; nurse; prevention
MeSH Terms: conditions — Pressure Ulcer | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Patients assigned to the experimental group will first be informed about the study by phone and their participation status will be questioned. The relatives of the patients who want to participate in the study will be visited at home with the Home Health Services unit of Izmir Atatürk Training and Research Hospital and the data collection process and training will be carried out. After the training is given, the caregiver will be questioned about the applicability of the training content and the need for reminder training by calling the caregiver weekly in the first month and every two weeks in the second and third months for three months, and will be evaluated in terms of pressure sore formation, primarily in risky areas, during these interviews or by using the records of home health services.
  Interventions: Other: education
- control group (No Intervention): Patients assigned to the control group must be home care patients who have registered with Izmir Atatürk Training and Research Hospital Home Health Services Unit within the last month, be over 18 years of age, be bedridden, and not have developed pressure sores on any part of their body. The caregivers of the patients assigned to the control group will be invited to the study by calling by phone, the introductory characteristics of the relatives of the patients who want to participate will be taken first, and the formation of pressure ulcers at the end of the first, second and third month without any training will be evaluated by calling by phone or by using the records of the Home Health Services Unit. At the end of the study, the patient / patient relatives assigned to the control group will also be given training to prevent pressure sores and a brochure will be given.

INTERVENTIONS:
Other: education — Prepared in clear language and supported with visuals in line with guidelines and studies (Kottner et al. 2019, Orhan 2017, APUPA 2011, EPUAP and NPUAP 2009, EPUAP 2019, Arıkan and vanGiersbergen 2019, Arslantaş et al. 2018) training will be given to prevent pressure ulcers. Training content will be sent to expert opinion for content validity. In the content of the training, the definition of pressure ulcers, how they develop, high-risk areas for wound formation, identification of risks, evaluation of the skin, skin care, lying positions and position changes, supporting bone protrusions with pillows, lying on a support surface, nutritional status and content, fluid intake will be discussed.
  Arms: experimental group

SUMMARY:
Pressure ulcers are wounds that typically occur on bony prominences, primarily due to external factors such as pressure, friction, and shear, as well as internal factors related to the patient. These ulcers can lead to serious health issues and have a high incidence rate, negatively impacting patients' quality of life, increasing hospitalization duration, and adding to healthcare costs. Prevention of pressure ulcers is considered an important indicator of care quality worldwide and in our country. International guidelines emphasize key points for preventing pressure ulcers, including risk assessment, skin assessment and care, nutrition, repositioning, support surface use, documentation, and education.

DETAILED DESCRIPTION:
A pressure ulcer is defined as "localized skin and/or subcutaneous tissue damage caused by pressure alone or in combination with pressure or tearing, usually occurring on bony prominences". Mostly, it develops as a result of prolonged compression of soft tissue between the bony prominence and the outer surface. External factors such as a large force applied for a short period of time or less force applied for a long period of time, friction, tearing, and stretching to which the skin is exposed disrupt the blood flow to the area, prevent oxygen and nutrient transport to the tissues and cause pressure sores. An overly moist environment caused by sweating, urinary or fecal incontinence or excessive wound drainage increases the harmful effects of pressure, friction and shearing. It also causes maceration of the surrounding skin, which combines these factors. Friction and moisture have their greatest effect in areas of high pressure. If moisture is present, the effects of friction increase up to five times. In addition, intrinsic risk factors associated with the development of pressure sores include old age (70 years and older), immobility/impaired mobility, dehydration, impaired sensory perception and tissue perfusion, malnutrition, anemia, low albumin levels, hypothermia, hypotensive episodes, diabetes and peripheral vascular disease, medications that cause vasoconstriction, current smoking history, dry skin, low Body Mass Index, altered mental status (e.g. confusion), urinary and fecal incontinence, physical limitations, malignancy, history of pressure ulcers. Urinary and fecal incontinence, physical limitations, malignancy, history of pressure ulcers. Pressure ulcers, a pathology with high morbidity and mortality, cause a significant increase in caregiver burden and care costs. Treatment of pressure sores ranks third in terms of cost after malignancies and cardiovascular diseases. In a study conducted in nursing homes in the UK, pressure ulcer treatment costs 1.4-2.1 billion pounds per patient. In Turkey, the annual cost is estimated to be $1 billion 425 million. The European Pressure Ulcer Advisory Panel (EPUAP) recommends that identifying pressure ulcers at Stage 1 and preventing complications and deepening by taking effective measures is the most effective way to reduce costs.

Today, guidelines have been developed in the light of evidence-based practices to prevent pressure ulcers. The main prevention interventions included in these guidelines are assessment of pressure ulcer risk, skin assessment and care, assessment and support of nutritional status, changing position, use of support surfaces, education of healthcare professionals, patients and their relatives, and record keeping. The simplest and easiest way to prevent the development of pressure sores is to take prevention measures. The basic approach in the prevention of pressure sores is to evaluate the possible risks to prevent the development of the wound before it occurs, early identification of the risk group and early implementation of prevention initiatives. EPUAP and NPUAP recommend that all bedridden patients with limited mobility should be considered in the risk group. In the light of all this information, in this study, it was aimed to provide training to the caregivers of bedridden patients to prevent pressure ulcers at home in line with the recommendation of the guidelines as one of the effective interventions in the prevention of pressure sores and to examine the effect of this training on pressure ulcer formation.

ELIGIBILITY:
Inclusion Criteria:

* Being a home care patient who has registered to Izmir Atatürk Training and Research Hospital Home Health Services Unit within the last month
* Being over 18 years of age
* Being bedridden
* Not having pressure sores on any part of the body

Exclusion Criteria:

* Patients who died during the data collection and follow-up process
* Changed their home/changed caregivers and/or did not speak Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
occurrence of pressure injury | 3 months
  Patients will be evaluated for pressure ulcers three months after the end of the training. In patients with pressure ulcers, the site and stage of the wound will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Ataturk Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No